CLINICAL TRIAL: NCT01638793
Title: Capnographic Monitoring of Propofol-sedation During Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: JWGUHMED1-006
Record Dates: First submitted 2012-07-11; First posted 2012-07-12 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2012-06

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Capnography (Experimental): Capnographic respiration monitoring
  Interventions: Device: Microcap (Oridion, Needham, MA, USA)
- Pulse-Oxymetry (Active Comparator): pulse-oxymetric respiration monitoring
  Interventions: Device: Smart Capno Line Plus O2 (Oridion, Needham, MA, USA)

INTERVENTIONS:
Device: Microcap (Oridion, Needham, MA, USA)
  Arms: Capnography
Device: Smart Capno Line Plus O2 (Oridion, Needham, MA, USA)
  Arms: Pulse-Oxymetry

SUMMARY:
The present study is a randomized, prospective, single-blinded study. Patients presenting for colonoscopy under sedation will be included according to the statistical sample size calculation. Patients will be randomized to either group 1- capnographic monitoring or group 2- oxygenic monitoring during Propofol-based sedation for colonoscopy. Episodes of Hypoxia are documented and compared in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Indication for colonoscopy
* Patient wishing sedation during colonoscopy
* ≥ 18 years of age
* Signed informed consent form

Exclusion Criteria:

* Diseases which preclude study accomplishment or put the patient at any risk (e.g. psychiatric diseases)
* Non-contractually capable persons
* Pregnancy
* Lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Hypoxia (SO2 <90%)
  Study objective is to evaluate if a reduction of hypoxic events (SO2 <90% for ≥ 15 sec) can be obtained with capnographic monitoring as compared to standard monitoring of respiration with pulse-oxymetry in patients receiving colonoscopy under Propofol-based sedation

SECONDARY OUTCOMES:
Severe Hypoxia (SO2 <85%)
  Evaluate events of severe hypoxia (SO2 < 85%) in group 1 (capnographic monitoring) as compared to group 2 (oxymetric monitoring)
Time to hypoxia
  Evaluate the time difference between abnormal ventilation shown on capnography machine and hypoxemia.
Hypoxia in relation to sedation
  Compare events of hypoxemia and severe hypoxemia during sedation with propofol only as compared to propofol/ketamin combination sedation.
Vegetative Symptoms
  Evaluate vegetative events (hypotension, hypertension, bradycardia, tachycardia, tachypnea, bradypnea) in both groups during the two sedation forms

CONTACTS AND LOCATIONS:
Overall Officials: Mireen Friedrich-Rust, MD, Principal Investigator — Klinikum der J. W. Goethe-Universität Frankfurt am Main
Locations (2):
- Germany (2):
  - Klinikum der J. W. Goethe-Universität, Frankfurt am Main
  - Praxisklinik am Staedel, Frankfurt am Main